CLINICAL TRIAL: NCT04510350
Title: Investigation of Novel Immunological Biomarkers by Mass Cytometry in Patients With Early Multiple Sclerosis (CISCO)
Acronym: CISCO
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_8880_CISCO
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS CIS+
  Interventions: Other: Biomarkers analysis
- Healthy volunteers
  Interventions: Other: Biomarkers analysis

INTERVENTIONS:
Other: Biomarkers analysis — Genetic analysis of regions of interest

SUMMARY:
The objective of CISCO is therefore to identify prognostic biomarkers of MS activity in early-stage patients.

ELIGIBILITY:
Patients :

Inclusion Criteria:

* Patients with clinically isolated syndrome (CIS) participating in the OFSEP cohort (French MS Observatory)
* At least 18 years of age
* Diagnosed with MS according to criteria 2017 at the time of their last visit.
* Non-opposition to participation in the study
* Having had at least one visit in the year following collection
* Follow-up for at least 1 year after collection.
* Having signed the OFSEP consent

Exclusion Criteria:

* CIS patients with progressive MS

Healthy volunteers :

Inclusion Criteria:

* Age 18 years or older
* Having participated in the ABCD-SEP clinical trial promoted by the Rennes University Hospital (NCT03744351).
* Matched on age and sex to patients of interest in the OFSEP cohort
* Not having objected to participation in the study

Exclusion Criteria:

* Persons of full age subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After selection of the patients and volunteers of interest (number and type of clinical and biological data available, heterogeneity of the chosen group...), the medical and imaging data of the patients will be transmitted by OFSEP from the EDMUS database and for healthy volunteers, the data of interest will be retrieved from the ABCD-SEP database
  Patients CIS+ :60 Healthy Volunters : 30
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Frequency of immune subpopulations | 1 year
  Correlations between the frequency of immune subpopulations, genetic profile and disease activity

SECONDARY OUTCOMES:
Frequency of immune subpopulations correlated to EDSS score | 1 year
  Correlations between the frequency of immune subpopulations, genetic profile, and EDSS score ((Expanded Disability Status Scale, method of quantifying disability in multiple sclerosis, steps 1.0 to 4.5 refer to people with MS who are fully ambulatory. EDSS steps 5.0 to 9.5 are defined by the impairment to ambulation.)
Frequency of immune subpopulations correlated to disease progression delay | 1 year
  Correlations between the frequency of immune subpopulations, genetic profile, and delay before disease progression
Frequency of immune subpopulations correlated to disease progression events | 1 year
  Correlations between the frequency of immune subpopulations, genetic profile, and number of disease progression events
Frequency of immune subpopulations correlated to spinal lesions | 1 year
  Correlations between the frequency of immune subpopulations, genetic profile, and number of new spinal lesions
Profiles of CIS+ patients | 1 year
  Comparison of genetic and immunological profiles of CIS+ patients with healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Laure Michel, Md, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided